CLINICAL TRIAL: NCT00717080
Title: Role of Capsular Tension Ring in Anterior Capsular Contraction in Retinitis Pigmentosa Patients
Brief Title: The Role of Capsular Tension Ring (CTR) in Anterior Capsular Contraction
Acronym: ACO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aurolab (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2PR1210826
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2009-10

CONDITIONS: Retinitis Pigmentosa; Cataract
Keywords: Retinitis Pigmentosa; Cataract
MeSH Terms: conditions — Retinitis Pigmentosa; Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): IOL surgery with Capsular Tension Ring
  Interventions: Procedure: IOL surgery
- Arm 2 (Placebo Comparator): IOL surgery without Capsular Tension Ring
  Interventions: Procedure: IOL surgery

INTERVENTIONS:
Procedure: IOL surgery — IOL surgery using capsular tension ring (AURORING)
  Other Names: AURORING
  Arms: Arm 1
Procedure: IOL surgery — IOL surgery without CTR
  Other Names: Phacoemulsification
  Arms: Arm 2

SUMMARY:
This is a Randomized Controlled Trial to study the role of Capsular Tension Ring in patients with Retinitis Pigmentosa

DETAILED DESCRIPTION:
Cataract is a common complication in retinitis Pigmentosa (RP) patient especially posterior sub capsular cataract. Continuous curvilinear capsulorhexis is the preferred method of capsulotomy in cataract surgery. Anterior capsular contraction (ACO) is a unique complication following cataract surgery. The rate of which is higher in RP patients due to the weak zonules and the increased rate of inflammation. CTR has been proven to reduce the rate of contraction.

Study population includes 40 eyes having RP with cataract. 20 eyes will receive CTR and the other 20 would not receive CTR. The percentage of anterior capsular contraction would be evaluated using EPCO software.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 65 years
* Typical retinitis pigmentosa
* Reside within a radius of 100kms from Madurai
* Patients willing to come for follow up
* Patients with nuclear sclerosis grade 2 or 3 or cortical cataract or pscc

Exclusion Criteria:

* Diabetic patients
* Traumatic cataract
* Uveitis
* Glaucoma
* Pseudoexfoliation
* Myotonic dystrophy
* Corneal pathology
* Pupil size <6mm
* Intra op complications like zonular dialysis,pc rupture
* Rhexis not covering iol optic

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The percentage of anterior capsular contraction | 1 day, 30 days,90 days,180 days,270days

SECONDARY OUTCOMES:
Visual acuity | 1 day, 30 days,90 days,180 days,270days

CONTACTS AND LOCATIONS:
Overall Officials: Haripriya Aravind, MS, Principal Investigator — Aravind Eye Hospital, Madurai
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India